CLINICAL TRIAL: NCT00310609
Title: Multicenter, Open-label Study of the Safety (Open-label) and Efficacy (Open-label and Blinded Reader) of a Single Administration of Approximately 0.1 mmol/kg of Magnevist® Injection-enhanced Magnetic Resonance Arteriography (MRA) and 2-dimensional-time-of-flight (2D-TOF) MRA in Patients With Known or Suspected Disease of the Aortic Arch and Cerebral Branches Who Are Undergoing MRA of These Vessels With Intra-arterial Digital Subtraction Arteriography (i.a. DSA) as the Standard of Reference.
Brief Title: Magnevist® Injection Enhanced MRA Compared to Non Contrast MRA for the Detection of Structural Abnormalities of the Aortic Arch and Cerebral Branches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90941; 304630
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Abnormalities
Keywords: Structural abnormalities of the aortic arch and cerebral branches
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist) — Gadopentetate dimeglumine (Magnevist Injection), approximately 0.1mmol/kg body weight, single intravenous administration on the study day

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Magnevist (the study drug) used for MRI of the aortic arch and cerebral branches. The results will be compared to the results of MRI taken without Magnevist, and with the results of your X-ray angiography.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has known or suspected disease of the aortic arch and cerebral branches
* Is scheduled for X-ray angiography

Exclusion Criteria:

* Has any contraindication to magnetic resonance imaging
* Is scheduled for any procedure before the X-ray angiography
* Had previous bilateral intervention (surgery, bypass) of the arteries of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2003-12; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Accuracy, sensitivity, and specificity based on quantitative assessment of stenosis assesses by blinded reader | Image creation after injection -evaluation at blind read

SECONDARY OUTCOMES:
Diagnostic confidence | At blinded and/or open label read of the images
Visual assessment of stenosis | At blinded and/or open label read of the images
Difference in degree of stenosis | At blinded and/or open label read of the images
Other diagnostic findings | At blinded and/or open label read of the images
Location and matching of stenosis | At blinded and/or open label read of the images
Image quality | At blinded and/or open label read of the images
Image evaluability and presence of artifacts | At blinded and/or open label read of the images
Ability to visualize arterial segments | At blinded and/or open label read of the images
Proportion of correctly categorized maximum stenosis per segment | At blinded and/or open label read of the images
Number of evaluable segments | At blinded and/or open label read of the images
Duration if 2D TOF and CE-MRA | At blinded and/or open label read of the images
Patient management | From baseline to 24 hours follow-up
Safety variables | From baseline to 24 hours follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer